CLINICAL TRIAL: NCT05382273
Title: Cannabis Tolerance Break Resource Study: T-Break Guide
Status: Completed | Type: Observational
Sponsor: University of Vermont (Other)
Collaborators: Dartmouth College (Other); Rutgers University (Other)
Responsible Party: Principal Investigator, Tom Fontana, Alcohol, Cannabis & Other Drugs Initiatives Manager, University of Vermont
Other Study IDs: STUDY00001489; 03420-08153 (Other Grant/Funding Number: State of Vermont - ADAP)
Record Dates: First submitted 2022-05-11; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Cannabis Use; Tolerance; Cannabis Withdrawal
Keywords: Open Pilot Study; Pre test / Post test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Use of T-Break Guide: None: Participants who reported not using the T-Break Guide (intervention)
- Use of T-Break Guide: Some: Participants who reported using the T-Break Guide "some"
  Interventions: Behavioral: T-Break Guide
- Use of T-Break Guide: A lot: Participants who reported using the T-Break Guide "a lot"
  Interventions: Behavioral: T-Break Guide

INTERVENTIONS:
Behavioral: T-Break Guide — The T-Break Guide was designed to help people complete a 21-day break from cannabis. For each day of the break, the Guide offers inspiration in the form of a quote, reflections based on likely experiences occurring at that point during the break, advice on ways to overcome challenges, alternative activities in which to engage, and encouragement.
  * The first week focuses on physical symptoms of cannabis withdrawal (e.g., sleep, appetite).
  * The second week focuses on the emotional experience (e.g., anxiety, boredom).
  * The third week focuses on behavioral aspects (e.g., examining patterns, connections).
  The T-Break Guide follows the Motivational Interviewing principles of affirmation and autonomy.
  Groups: Use of T-Break Guide: A lot; Use of T-Break Guide: Some

SUMMARY:
The purpose of this pilot study is to conduct research into the value of using the T-Break Guide for assisting people taking a tolerance break from cannabis. The hope is that this initial research will yield some insights and benchmarks into the Guide's efficacy, and provide a foundation for a later randomized control study.

The following are some key research questions:

1. How did participants use the Guide? (Eg: daily; read once; 'a la carte')
2. How did using the Guide increase fidelity to tolerance break (starting, continuing, completing a break)?
3. Did using the Guide yield any benefits beyond tolerance break fidelity? (Eg: insight into patterns of use)

DETAILED DESCRIPTION:
The pilot study used a pretest-posttest design in which participants completed a baseline survey and were asked to attempt a 21-day period of cannabis abstinence, to consider using the T-Break Guide (intervention) in their attempt, and to complete a follow-up survey after 30 days.

Participants were young adults aged 18-29 recruited through posters and tabling events at the University of Vermont (UVM), a post on a UVM webpage, emails on listservs of seven other universities, and a post on a subreddit focusing on responsible cannabis use. The posters and online announcements directed participants to the online baseline survey, which contained consent information before allowing participants to complete.

After completing the baseline survey, participants received a link to an online version of the T-Break Guide through email. After 30 days, participants received another email prompting them to complete the follow-up survey. The UVM Institutional Review Board reviewed and approved all study procedures (STUDY00001489).

ELIGIBILITY:
Inclusion Criteria:

* Current cannabis partakers, willing to attempt at 21 day tolerance break (ie, period of cannabis abstinence)

Exclusion Criteria:

* No cannabis use in past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants were young adults aged 18-29 recruited through posters and tabling events at the University of Vermont (UVM), a post on a UVM webpage, emails on listservs of seven other universities, and a post on a subreddit focusing on responsible cannabis use. The posters and online announcements directed participants to the online baseline survey, which contained consent information before allowing participants to complete.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Tolerance Break Completion | 21 days
  Did the participant go 21 days without using cannabis? Self-report, "yes/no" question on followup survey

SECONDARY OUTCOMES:
Cannabis Use After 21 Days | 21 days
  How much cannabis are participants using after 21 days break? Followup survey question, 5 point Likert scale with "way more; a little more; same; a little less; way less" as response options
Confidence in Future Break | 30 days
  Participants' confidence level about how successful they would be taking a future break
Important of Balance | 30 days
  Participants' importance with finding/keeping balance in cannabis use going forward
Alcohol and Other Drug Use During Break | 30 days
  What happened to participants' alcohol and other drug use while stopping cannabis? Self report by category of substance, asking use prior and change (if any) during break
Future Cannabis Use | 30 days
  After taking a break, where do participants' picture their cannabis use in 3 years? Followup survey question, "Where do you picture your cannabis use 3 years from now" {"a lot more; a little more; about the same; a little less; a lot less; none}

CONTACTS AND LOCATIONS:
Overall Officials: Tom Fontana, MS, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Yes
Non identifiable participant data is planned to be shared via a free data repository
Access Criteria: Free and open

REFERENCES:
- [Background] Enkema MC, Hallgren KA, Larimer ME. Craving is impermanent and it matters: Investigating craving and cannabis use among young adults with problematic use interested in reducing use. Drug Alcohol Depend. 2020 May 1;210:107957. doi: 10.1016/j.drugalcdep.2020.107957. Epub 2020 Mar 14. PMID 32200158
- [Background] Enkema MC, Hallgren KA, Bowen S, Lee CM, Larimer ME. Craving management: Exploring factors that influence momentary craving-related risk of cannabis use among young adults. Addict Behav. 2021 Apr;115:106750. doi: 10.1016/j.addbeh.2020.106750. Epub 2020 Dec 3. PMID 33383565
- [Background] Schuster RM, Gilman J, Schoenfeld D, Evenden J, Hareli M, Ulysse C, Nip E, Hanly A, Zhang H, Evins AE. One Month of Cannabis Abstinence in Adolescents and Young Adults Is Associated With Improved Memory. J Clin Psychiatry. 2018 Oct 30;79(6):17m11977. doi: 10.4088/JCP.17m11977. PMID 30408351